CLINICAL TRIAL: NCT04202900
Title: Exploring the Effectiveness of LED Phototherapy on Common Symptoms Among Elderly in Long-Term Care Institutions and Its Translation Application
Brief Title: Exploring the Effectiveness of LED Phototherapy on Common Symptoms Among Elderly in Long-Term Care Institutions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: YM108088E
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Low Level Light Therapy
Keywords: elderly; LED phototherapy; meridian energy; sleep quality; fatigue; cold limbs; long-term care institution
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phototherapy protocol (Other): Pretest：Common symptoms in the elderly include insomnia, depression, pressure sore wounds, blood sugar, blood pressure, body temperature,fatigue,cold limbs.
  Intervention：LED light therapy for 6 weeks, 2-3 times a week, every 30 minutes. Post test：Common symptoms in the elderly include insomnia, depression, pressure sore wounds, blood sugar, blood pressure, body temperature,fatigue,cold limbs.
  Interventions: Other: phototherapy protocol

INTERVENTIONS:
Other: phototherapy protocol — Pretest：Common symptoms in the elderly include insomnia, depression, pressure sore wounds, blood sugar, blood pressure, body temperature,fatigue,cold limbs.
  Intervention：LED light therapy for 6 weeks, 2-3 times a week, every 30 minutes. Post test：Common symptoms in the elderly include insomnia, depression, pressure sore wounds, blood sugar, blood pressure, body temperature,fatigue,cold limbs.

SUMMARY:
The world is facing rapid population aging, the health needs of the elderly are complex, and their physical capabilities are degraded, and increased the possibility of having one or more chronic conditions. In 1900 to 2000, there were 7,600 million people in the United States, aged 65 and above age increased to 4.1% up to 12.6%, by 2050 is expected to increase 20.3%.In Taiwan, the elderly population have 83.5% is health and sub-health, in order to allow them to perform activities of daily living independently, in particular, need to pay attention to the diverse needs of the elderly, Assist the elderly to increase self-care skills, reduce disability is a very important issue.

DETAILED DESCRIPTION:
From literature review of LED phototherapy can effectively improve symptoms in the elderly, such as hair loss, dermatitis, rotator tendonitis, epicondylitis of the tibia, wound healing, back pain, patellofemoral pain, spinal neuropathy, chronic pain relief, insomnia and depression.

Comprehensive Phototherapy and Traditional Chinese medicine(TCM) perspective, LED phototherapy is the use of physical light energy stimulation and temperature to improve the body's microcirculation and meridian dredge, Enhance the body's energy of the health and sub-health elderly, increasing physical activity perform daily functions.

Taiwanese Elderly to take self-care by the dilemmas of the many aspects. There are 21.52% physical health problems, affecting work or daily activities are limited; there are 35.12% physical or emotional health problems affecting social activities; there are 13.01% incapable perform activities of daily living.

The aim of this study was to explore the effectiveness of LED phototherapy on physiological symptoms among elderly in long-term care institutions in Taiwan. To examine the effects of physiological symptoms, such as mental state, muscle bone system, metabolism, autonomic balance and other meridian energy tests, it is expected to improve the body energy of healthy and sub-healthy elderly to increasing physical activity perform daily functions.

ELIGIBILITY:
Inclusion Criteria:

* Consciousness clear；must be able to talk

Exclusion Criteria:

* Clinical diagnosis of dementia；Seasonal mood disorder

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index/PSQI | Change before, through intervention completion (average 6 weeks).
  Insomnia was measured by the Pittsburgh Sleep Quality Index (PSQI), Global PSQI >5 score，good sleep；Global PSQI ≦5 score，poor sleep。
Brief Fatigue Inventory-Taiwanese (BFI-T) | Change before, through intervention completion (average 6 weeks).
  Fatigue was measured by the Brief Fatigue Inventory-Taiwanese (BFI-T), BFI-T=0 score，no fatigue；1~3 score，A little tired (not tired most of the time)；4~6 score，Ordinary tired, tolerable (about half the time to feel tired)；7~9 score，very tired (most of the time feel tired)；10 score，most tired (I feel tired all the time)。
Cold Limbs | Change before, through intervention completion (average 6 weeks).
  Cold Limbs was measured by the Yes / No Questionnaire elderly subjective feeling, "Yes" in the questionnaire means cold limbs；"No" in the questionnaire means no cold limbs。
Braden-Pressure ulcer risk factor assessment scale | Change before, through intervention completion (average 6 weeks).
  Pressure ulcer was measured by the Braden-Pressure ulcer risk factor assessment scale, ≧16 score，Low-risk；12-15 score，Moderate risk；≦11 score，High-risk。

SECONDARY OUTCOMES:
Meridian Energy | Measured 1 week before and 1, 4, 6 weeks after intervention
  Meridian energy was examined by using the Meridian Energy Analysis Device(M.E.A.D.), Parameters and normal values：Mental health status：0.78-1.09；Musculoskeletal status：0.88-1.14；Metabolism status：0.82-1.24；Autonomic nervous system status：1.0-1.5；Overall energy：28-64。
HRV | Measured 1 week before and 1, 4, 6 weeks after intervention
  Autonomic nervous system activity was examined by using the Heart Rate Variability (HRV), Parameters and normal values：Low Frequency power(LF)：0.04~0.15 Hz；High Frequency power(HF)：0.15~-0.4 Hz；Standard deviation(SD)：All normal to normal intervals, the larger the SD, the greater the HRV；mean Heart Rate；LF/HF ratio。
Body Temperature | Measured 1 week before and 1, 4, 6 weeks after intervention
  Cold Limbs was measured by the body temperature (BT), Ear temperature measurement normal BT 36 ~ 37.5。

CONTACTS AND LOCATIONS:
Locations (1):
- Chong-En Group Long-term Care Center for the Elderly, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No